CLINICAL TRIAL: NCT01441518
Title: A Prospective Randomized Trial of Home Versus Hospital Care in Glucose Monitoring of Gestational Diabetes and Mild Gestational Hyperglycemia
Brief Title: Home Versus Hospital Care in Glucose Monitoring of Gestational Diabetes and Mild Gestational Hyperglycemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Silvana Andrea Molina Lima, PhD, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-52
Record Dates: First submitted 2011-05-31; First posted 2011-09-27 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2011-09

CONDITIONS: Gestational Diabetes Mellitus; Pregestational Diabetes Mellitus; Mild Gestational Hyperglycemia
MeSH Terms: conditions — Diabetes, Gestational | interventions — Home Care Services

ARMS (2):
- Home care (Experimental)
  Interventions: Other: Home care
- Hospital care (Active Comparator)
  Interventions: Other: Hospital care

INTERVENTIONS:
Other: Home care — Home care, sometimes called "ambulatory care" or "outpatient", was defined as the blood-glucose self-monitored by the pregnant women at home. This project will provide glucometers to all those who are randomized to home care. The women will receive training for glucose control in pre-defined days, with the glucometer to obtain the mean glucose. According to blood-glucose levels in glycemic profile, insulin dose will be maintained or altered both in gestational diabetes as in mild gestational hyperglycemia .
  Arms: Home care
Other: Hospital care — Hospital care, sometimes called "acute care", was defined as control of maternal diabetes made at hospitals by admission to hospital. The blood-glucose and metabolic control are done in gestational diabetes and mild gestational hyperglycemia treated conventionally.
  The hospitalized patients will have their glycemic control done in the hospital. . According to blood-glucose levels in glycemic profile , insulin dose will be maintained or altered both in gestational diabetes as in mild gestational hyperglycemia.
  All the women of the study will be accompanied by a team of obstetricians specializing in high-risk pregnancies; residents; dietitians; nurses and neonatologists.
  Arms: Hospital care

SUMMARY:
Pregnancies complicated by diabetes and mild gestational hyperglycemia are associated with increased perinatal and maternal complications. The most serious maternal complication is the risk of developing type 2 diabetes after 10-12 years of the delivery. Perinatal complications include fetal macrosomia with consequent increased risk of obstetrical trauma and hypoxia/asphyxia, high rates of cesarean section, respiratory distress syndrome, and metabolic disorders at birth. Regardless of the diagnosis of diabetes and mild gestational hyperglycemia, the perinatal outcome is directly related to maternal metabolic control. For the tight control of blood glucose, pregnant women are treated as home care (outpatient) or hospital care. Objective: To evaluate the cost-effectiveness and safety of home versus hospital care of gestational diabetes and mild gestational hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with gestational, pre gestational diabetes mellitus or mild gestational hyperglycemia. Patients should have one of the four criteria as following:
* Patients with positive screening for GDM presenting a TTG of 75 g and one of the values below:

  * fasting glucose ≥ 92;
  * 1h ≥ 180; or
  * 2h ≥ 153 will be considered gestational diabetes mellitus (GDM) and these patients will be enrolled to a run-in phase consisting of diet and exercise during 15 days. If the patients still present an abnormal glycemic profile instead of the previous treatment with diet and exercise they will be enrolled in the study and randomized to either home or hospital care; or
* Patients with pre gestational diabetes mellitus type 1 or 2; or
* Patients with positive screening for GDM and presenting normal TTG of 75 g and abnormal glycemic profile, fasting ≥ 85 mg k/l 10 h to 18h post prandial ≥ 130 mg k/ ( Rudge et al,1990).
* Normal TTG and an abnormal glycemic profile will be considered as mild gestational hyperglycemia
* Patient provided written informed consent.

Exclusion Criteria:

* Twin pregnancy diagnosed until the date of randomization or;
* Fetal malformation diagnosed until the date of randomization.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maternal mortality and morbidity rates | participants will be followed regarding maternal and perinatal mortality and morbidity rates up to six weeks postnatal
Perinatal mortality and morbidity rates | participants will be followed regarding maternal and perinatal mortality and morbidity rates up to six weeks postnatal

SECONDARY OUTCOMES:
Birth weight (classified as appropriate for gestational age = AIG, small for gestational age =SGA and large for gestational age = LGA) | birth weight will be assessed for an expected average of 9 months from the time of randomization
Maternal hospitalizations for any causes (home care) and prolonged hospitalization (hospital care) | participants will be followed for maternal hospitalizations for any causes and prolonged hospitalization up to six weeks postnatal
Infants repeated hospitalizations | infants will be followed for repeated hospitalizations up to six weeks postnatal
Infants acute care visits | infants will be followed for acute care visits up to six weeks postnatal
Length of stay for delivery | participants will be followed for length of stay for delivery, an expected average of 9 months
Maternal prenatal and postpartum acute care visits | participants will be followed for maternal prenatal and postpartum acute care visits up to six weeks postnatal
Biophysical profile tests | participants will be followed for biophysical profile tests up to six weeks postnatal
Incidence of premature infants | participants will be followed regarding incidence of premature infants up to six weeks postnatal
Postpartum repeated hospitalization | participants will be followed for Postpartum repeated hospitalization up to six weeks postnatal
Glucose control | participants will be followed for glucose control up to six weeks postnatal
Costs | costs will be assessed for an expected average of 9 months from the time of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Dr Regina El Dib, PhD, Study Director — UPECLIN HC FM Botucatu Unesp; Dr Marilza Rudge, PhD, Principal Investigator — UPECLIN HC FM Botucatu Unesp
Locations (1):
- Faculdade de Medicina de Botucatu, Universidade Estadual Paulista, Botucatu, São Paulo, Brazil